CLINICAL TRIAL: NCT00761423
Title: The Value of Platelet-Rich Plasma in Chronic Midportion Achilles Tendinopathy: a Double-blind Randomized Clinical Trial
Acronym: PRICT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMET NL 02; NTR1420
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Achilles Tendinopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Combination of eccentric exercises and injection of PRP
  Interventions: Biological: PRP Injection with eccentric exercises
- 2 (Placebo Comparator): Combination of eccentric exercises and physiological saline injection
  Interventions: Biological: Placebo Injection with eccentric exercises

INTERVENTIONS:
Biological: PRP Injection with eccentric exercises — PRP Injection with eccentric exercises
  Arms: 1
Biological: Placebo Injection with eccentric exercises — Placebo Injection with eccentric exercises
  Arms: 2

SUMMARY:
The study will be a double-blind randomized single-center clinical trial comparing 3 treatment groups with chronic midportion Achilles tendinopathy.

DETAILED DESCRIPTION:
Introduction- Overuse injury of the Achilles tendon is a common entity in athletes and older athletes are at an increased risk. When the exact origin of tendon pain is unclear, the term tendinopathy is preferred. Most accepted treatment at this moment is an eccentric exercise programme, according to the Dutch guidelines. However, a recent systematic review on the effectiveness of eccentric exercises to treat lower extremity tendinoses concluded that it is unclear whether eccentric exercises are more effective than other forms of treatment.

Recent studies described new treatment strategies in tendinopathies, such as the use of platelet-rich plasma (PRP). Platelets can participate actively in tissue repair processes and stimulate the release of several growth factors. Recently, it was found that platelet-rich plasma clot releasate stimulates cell proliferation, collagen deposition, and enhances the gene expression of matrix degrading enzymes and endogenous growth factors by human tendon cells in vitro. The only published clinical cohort study in tendon research reported 93% reduction of pain for PRP-treated patients with chronic elbow tendinosis. Also on short term follow-up, the PRP injection was more beneficial than injection with an anaesthetic agent.

Aim- To monitor the potential clinical improvement of chronic midportion Achilles tendinopathy after injection with PRP and to evaluate the recovery process in time using a new Ultrasonographic method (Ultrasonographic Tissue Characterisation).

Hypothesis: The average VISA-A score is higher in the patient group treated with eccentric exercise therapy in combination with a PRP injection in comparison with the group treated with a saline injection in combination with eccentric exercises.

Study population- In total, 54 patients with symptomatic Achilles tendinopathy will be included in the study.

Study design- The study will be a double-blind randomised single-centre clinical trial comparing 2 treatment groups. The researcher, the sports medicine physician and the patients will be blinded to the received therapy.

Therapy- All patients will perform a heavy load eccentric exercise programme, consisting of 180 repetitions daily. The patients will be randomised into 2 treatment groups: ultrasound guided intratendinous saline injection with eccentric exercises and ultrasound guided intratendinous PRP injection with eccentric exercises.

Follow-up- Follow-up (clinically and ultrasonographically) will be at 6, 12, 24 and 52 weeks. At 24 weeks, the researcher will be unblinded after the analysis of the preliminary data. The patients will remain blinded to the therapy until 52 weeks follow-up. At 52 weeks follow-up a second, blinded researcher will evaluate the patients using the primary and secondary outcome measurements.

Outcome measurements- Primary outcome measurement: VISA-A score, a validated instrument to detect the severity of symptoms in patients with Achilles tendinopathy. As secondary outcome measurements subjective patient satisfaction and return to sports will be rated. For the evaluation of tendon repair, Ultrasonographic Tissue Characterization (UTC) and Power Doppler ultrasound (PDU) will be performed. UTC was previously developed in horse tendons and provides quantitative information on tendon fiber alignment and the related ultra-structural integrity of the tendon tissue through a non-invasive approach.

ELIGIBILITY:
Inclusion criteria

1. Clinical diagnosis "chronic midportion Achilles tendinopathy"
2. Age 18-70 years

Exclusion criteria

1. Clinical suspicion of insertional disorders (pain at the site of the insertion of the Achilles tendon on the calcaneum)
2. Clinical suspicion of an Achilles tendon rupture (Thompson test abnormal and palpabel "gap")
3. Clinical suspicion of plantar flexor tenosynovitis (posteromedial pain when the toes are plantar flexed against resistance)
4. Clinical suspicion of n.suralis pathology (sensitive disorder in the area of the sural nerve)
5. Clinical suspicion of peroneal subluxation (visible luxation of the mm. Peroneï spot in combination with localized pain)
6. Suspicion of internal disorders: spondylarthropathy, gout, hyperlipidemia, Rheumatoid Arthritis and sarcoidosis.
7. Condition that prevents the patients from executing an active exercise programme
8. Patient has already performed eccentric exercises, according to the schedule of Alfredson et al (12 weeks)
9. Patient has already received an injection of PRP for this injury
10. Patient does not wish, for whatever reason, to undergo one of the two treatments
11. Known presence of a pregnancy
12. Condition of the Achilles tendon caused by medications (arising in relation to moment of intake), such as quinolones and statins

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
VISA-A Score | 6, 12, 24 and 52 weeks

SECONDARY OUTCOMES:
Ultrasonographic Tissue Characterization | 6,12, 24 and 52 weeks
Complications | Anytime
Power doppler sound | 6, 12, 24 and 52 weeks
Patient satisfaction | 6, 12, 24 and 52 weeks
Return to sport | 6, 12, 24 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: RJ De Vos, MD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

REFERENCES:
- [Derived] Lagas IF, Tol JL, Weir A, de Jonge S, van Veldhoven PLJ, Bierma-Zeinstra SMA, Verhaar JAN, de Vos RJ. One fifth of patients with Achilles tendinopathy have symptoms after 10 years: A prospective cohort study. J Sports Sci. 2022 Nov;40(22):2475-2483. doi: 10.1080/02640414.2022.2163537. Epub 2023 Jan 8. PMID 36617848
- [Derived] de Vos RJ, Weir A, van Schie HT, Bierma-Zeinstra SM, Verhaar JA, Weinans H, Tol JL. Platelet-rich plasma injection for chronic Achilles tendinopathy: a randomized controlled trial. JAMA. 2010 Jan 13;303(2):144-9. doi: 10.1001/jama.2009.1986. PMID 20068208